CLINICAL TRIAL: NCT04857983
Title: Memantine Augmentation of Targeted Cognitive Training in Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Gregory Light, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201502
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; cognitive training; EEG
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to targeted cognitive training (TCT) and memantine (MEM) or targeted cognitive training (TCT) and placebo (PBO)
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized to TCT and memantine or TCT and placebo. The research will be provided with a randomization scheme to follow and will dispense the pills identified only by a code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TCT + PBO (Placebo Comparator): Subjects will be assigned to take placebo and will complete 30 hours of targeted cognitive training in order to assess whether memantine enhances cognitive training performance
  Interventions: Drug: Placebo
- TCT + MEM (Active Comparator): Subjects will be assigned to take memantine and will complete 30 hours of targeted cognitive training in order to assess whether memantine enhances cognitive training performance
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Subjects will be assigned to take memantine or placebo and will complete 30 hours of targeted cognitive training in order to assess whether memantine enhances cognitive training performance
  Other Names: targeted cognitive training (TCT)
  Arms: TCT + MEM
Drug: Placebo — Subjects will be assigned to take memantine or placebo and will complete 30 hours of targeted cognitive training in order to assess whether memantine enhances cognitive training performance
  Other Names: targeted cognitive training (TCT)
  Arms: TCT + PBO

SUMMARY:
Treatment of schizophrenia currently includes antipsychotic medications and cognitive therapies which improve some symptoms, but do not sufficiently restore cognitive functioning or reduce psychosocial disability. We hypothesize that medications that specifically target sensory information processing deficits, rather than psychotic symptoms per se, will significantly enhance the benefits of a sensory-based targeted cognitive training (TCT) intervention in patients with schizophrenia. We will complete a randomized, double-blind clinical trial to: 1) confirm that the drug memantine augments TCT learning; 2) determine whether memantine enhances the clinical benefits from a full 30 session course of TCT vs. TCT plus placebo in antipsychotic- medicated schizophrenia patients, and 3) determine if memantine's enhancement of TCT is most effective in biomarker-defined subgroups of patients.

DETAILED DESCRIPTION:
Treatment of schizophrenia (SZ) currently includes antipsychotic medications and cognitive therapies which improve some symptoms, but do not sufficiently restore cognitive functioning or reduce psychosocial disability. We propose and will test a novel "augmentation strategy" for using medications to specifically enhance the benefits of targeted cognitive training (TCT) in schizophrenia. This project tests a rational and empirically supported platform for augmenting the benefits of TCT in antipsychotic medicated SZ patients by adjunctive daily treatment of 20 mg memantine, an FDA approved medication for the treatment of cognitive dysfunction in Alzheimer's Disease. We hypothesize that medications that specifically target sensory information processing deficits, rather than psychotic symptoms per se, will significantly enhance the benefits of a sensory-based targeted cognitive training (TCT) intervention in patients with schizophrenia. We will complete a randomized, double-blind clinical trial to: 1) confirm that the drug memantine augments TCT learning; 2) determine whether memantine enhances the clinical benefits from a full 30 session course of TCT vs. TCT plus placebo in antipsychotic- medicated schizophrenia patients, and 3) determine if memantine's enhancement of TCT is most effective in biomarker-defined subgroups of patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Written informed consent to participate in the study
* Age 18-65
* Absence of dementia or mental retardation
* Urine toxicology negative for recreational drugs
* Fluent and literate in English

Exclusion Criteria:

* Meets DSM-IV criteria for current substance abuse or dependence and has been substance abstinent for less than 30 days
* A history of traumatic brain injury
* Auditory or visual impairments severe enough to prevent study participation
* Under conservatorship (determined by Anasazi)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Positive & Negative Symptom Scale total (PANSSt) | approximately 13 weeks
  PANSS Total Score is the primary clinical outcome measured at baseline vs. post TCT session 10, 20 and 30 (approximately 13 weeks). The PANSS total score has a range 30-210, with higher scores indicating worse outcome.
World Health Organization Disability Schedule (WHODAS 2.0) | approximately 13 weeks
  Function will be assessed via the World Health Organization Disability Schedule 2.0 (WHODAS 2.0) at baseline vs. post-TCT session 10, 20 and 30 (approximately 13 weeks). The World Health Organization Disability Schedule (WHODAS 2.0) has a range 12-60, with higher scores indicating worse outcome.
MATRICS Consensus Cognitive Battery Global Composite T-score (MCCB-C) | approximately 13 weeks
  The MCCB Global Composite T-score (MCCB-C) is the primary neurocognitive outcome measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 13 weeks). The MATRICS Consensus Cognitive Battery (MCCB) composite T-score has no minimum or maximum score because it uses T-scores, which are standardized based on a community sample. A normal range MCCB composite T-score is between 40 and 60 and higher scores indicate better neurocognitive outcome.

SECONDARY OUTCOMES:
Positive & Negative Symptom Scale (PANSS) - positive symptom subscale | approximately 13 weeks
  Positive & Negative Symptom Scale (PANSS) positive symptom subscale measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 13 weeks). The PANSS positive symptom subscale is rated from 1 to 7 points ranging from absent to extreme. The range for the Positive Symptom subscale is 7-49 and higher scores indicate worse outcome.
Positive & Negative Symptom Scale (PANSS) - negative symptom subscale | approximately 13 weeks
  Positive & Negative Symptom Scale (PANSS) negative symptom subscale measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 13 weeks). The PANSS negative symptom subscale is rated from 1 to 7 points ranging from absent to extreme. The range for the negative symptom subscale is 7-49 and higher scores indicate worse outcome.
Psychotic Symptoms - PSYRATS hallucination subscale | approximately 13 weeks
  Psychotic Symptom Rating Scales (PSYRATS hallucination subscale) measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 13 weeks). The PSYRATS auditory hallucinations subscale (AHS) consisting of 11 items, with each item being rated from 0 (absent) to 4 (severe), range 0-44, with higher scores indicating more severe auditory hallucinations or worse outcome.
Manic Symptoms - Young Mania Rating Scale | approximately 13 weeks
  Young Mania Rating Scale total score measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 13 weeks). The range for the YMRS total score is 0-60, with higher scores indicating more severe manic symptoms or worse outcome.
Current Depressive Symptoms - PHQ-9 | approximately 13 weeks
  Patient Health Questionnaire-9 (PHQ-9) total score measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 13 weeks). The PHQ-9 has a range from 0 to 27 with higher scores indicating more severe depression or worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Teaching Facility (CTF B-403 at UCSD Medical Center), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT04857983/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT04857983/ICF_000.pdf